CLINICAL TRIAL: NCT01166711
Title: SeQuent 1000 - Treatment of Coronary Artery Disease With Bare Metal Stent Followed by Paclitaxel-Coated Balloon Catheter Versus Paclitaxel-Eluting Stent: Randomized Trial
Brief Title: Treatment of Coronary Artery Disease (CAD) With Bare Metal Stent (BMS) Followed by Paclitaxel-Coated Balloon Catheter Versus Paclitaxel-Eluting Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEQUENT 1000
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bare Metal Stent (BMS) followed by Drug Eluting Balloon (DEB) (Experimental)
  Interventions: Device: Coroflex Blue (BMS) followed by SeQuent Please (DEB)
- Drug Eluting Stent (DES) (Active Comparator)
  Interventions: Device: Coroflex Please (DES)

INTERVENTIONS:
Device: Coroflex Blue (BMS) followed by SeQuent Please (DEB) — * standard techniques will be used
  * maximal vasodilatation after nitro application
  * baseline angiography with at least two orthogonal views (showing target lesion free of foreshortening or vessel overlap)
  * 6 French guiding catheter at least
  * target lesion will be crossed with standard guidewire
  * direct stenting at the discretion of the investigator
  * if pre-dilation, a commercially available balloon will be used (length not exceeding the stent to be implanted)
  * full lesion coverage will be ensured (with one or more stents)
  * only insert assigned stent type
  * BMS needs to be fully embedded in vessel wall
  * post-dilation with high pressure is required before treatment with DEB
  * DEB will be inflated with nominal pressure (balloon equates to vessel diameter)
  * length of DEB should exceed the BMS by 2-3 mm on each side
  * if dissection, full length of dissection and optional additional stented area should be treated with additional DEB (to avoid geographic miss)
  Other Names: Coroflex Blue; Cobalt Chromium stent; BMS; SeQuent Please; Paclitaxel-coated Balloon Catheter; DEB
  Arms: Bare Metal Stent (BMS) followed by Drug Eluting Balloon (DEB)
Device: Coroflex Please (DES) — * standard techniques will be used
  * maximal vasodilatation after nitro application
  * baseline angiography with at least two orthogonal views (showing target lesion free of foreshortening or vessel overlap)
  * 6 French guiding catheter at least
  * target lesion will be crossed with standard guidewire
  * direct stenting at the discretion of the investigator
  * if pre-dilation, a commercially available balloon will be used (length not exceeding the stent to be implanted)
  * full lesion coverage will be ensured (with one or more stents)
  * only insert assigned stent type
  Other Names: Coroflex Please; Paclitaxel-Eluting Stent; DES
  Arms: Drug Eluting Stent (DES)

SUMMARY:
The purpose of this study is to compare the one-time application of Paclitaxel from SeQuent Please (Paclitaxel-coated Balloon Catheter) after using the Coroflex Blue (Cobalt Chromium Stent) with the slow releasing of small dose of Paclitaxel from the Coroflex Please (Paclitaxel-Eluting Stent) stent system in a non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease including patients with chronic stable angina, unstable angina and silent ischemia
* Presence of one or more coronary artery stenosis >50% in a native coronary artery from 2.25 to 3.5 mm in diameter that can be covered with one stent
* One lesion treated with the study device

Exclusion Criteria:

* Pregnancy
* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, paclitaxel, cobalt, chromium or contrast material
* Inability to provide informed consent
* Currently participating in another trial before reaching the primary endpoint
* Elective surgery within 12 months of percutaneous coronary intervention (PCI) unless dual antiplatelet therapy is maintained throughout the peri-surgical period
* Acute or recent myocardial infarction
* left ventricular ejection fraction (LVEF) < 30 %
* Stroke or transient ischemic attack within 6 months
* Stented segment longer than 23 mm
* Vessel diameter of less than 2,5 mm
* Significant calcification, chronic total occlusion (CTO) or thrombus in the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) - target vessel failure (TVF) | 9 months
  consisting of the composite of cardiac death, myocardial infarction (Q-wave and Non-Q wave) localized at the territory supplied by the treated vessel or target vessel revascularization (TVR) by either percutaneous coronary intervention or bypass graft surgery in the overall population

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 year
  defined as the composite of cardiovascular death, stroke, myocardial infarction (MI) or ischemia-driven target lesion revascularization (TLR), as well as the individual components of target vessel revascularization (TVR) and Major adverse cardiac events (MACE) and stent thrombosis
in-stent binary restenosis | 9 months
  defined as >= 50 % diameter stenosis (% DS)
Angiographic and clinical stent thrombosis | 30 days
Angiographic and clinical stent thrombosis | 6 months
Angiographic and clinical stent thrombosis | 9 months
Angiographic and clinical stent thrombosis | 1 year
Angiographic and clinical stent thrombosis | 2 years
Angiographic and clinical stent thrombosis | 3 years
In-stent and in-segment minimal luminal diameter (MLD) | 9 months
In-segment percent diameter stenosis (%DS) | 9 months
In-stent and in-segment late luminal loss | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Paweł E. Buszman, MD, PhD, Principal Investigator — American Heart of Poland, Katowice
Locations (1):
- Upper Silesian Heart Center, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zurakowski A, Buszman PP, Milewski KP, Janas A, Gorycki B, Kondys M, Gasior P, Michalak M, Boxberger M, Peppas A, Granada JF, Buszman PE. Stenting and Adjunctive Delivery of Paclitaxel Via Balloon Coating Versus Durable Polymeric Matrix for De Novo Coronary Lesions: Clinical and Angiographic Results from the Prospective Randomized Trial. J Interv Cardiol. 2015 Aug;28(4):348-57. doi: 10.1111/joic.12210. PMID 26224390